CLINICAL TRIAL: NCT01659879
Title: Multimedia Based Information to Parents in a Pediatric Acute Ward: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LBK-2010/12-1
Record Dates: First submitted 2012-08-02; First posted 2012-08-08 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Health Communication
Keywords: Parents; Caregivers; Anxiety; Consumer satisfaction
MeSH Terms: conditions — Anxiety Disorders; Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- multimedia information (Experimental): Health information concerning the child's diagnosis, treatment and recovery time after evaluation by the pediatrician, using a 15 minutes long standardized health information package with multimedia elements from the Norwegian website www.syktbarn.no (English version: www.childhealthguide.com)
  Interventions: Behavioral: Multimedia information
- verbal information (Active Comparator): Verbal health information by a nurse in the acute ward concerning the child's diagnosis, treatment and recovery time, after the evaluation by the pediatrician
  Interventions: Behavioral: verbal information

INTERVENTIONS:
Behavioral: Multimedia information
  Arms: multimedia information
Behavioral: verbal information
  Arms: verbal information

SUMMARY:
The aim of this study is to determine whether multimedia based health information presented in a pediatric acute ward to parents of children with breathing difficulties due to lower respiratory tract infections, is more effective than verbal information to reduce the parent's anxiety and to increase satisfaction with nursing care and health information.

DETAILED DESCRIPTION:
The intervention website www.syktbarn.no is an open Norwegian online resource for parents of small children, and the site contains videos, audio clips, animations, illustrations, pictures and text materials regarding children's illnesses and normal development. In addition, the parents can use an interactive symptom checker that will help them to decide what to do and when to seek medical advice when their child is sick. The uniqueness of the website is the authentic video clips of sick children with common childhood symptoms like breathing difficulties, signs of dehydration, rash, cough and fever.

ELIGIBILITY:
Inclusion Criteria:

* parents of 0-15 years old children with breathing difficulties caused by LRTI (bronchiolitis, laryngitis or pneumonia) or asthma exacerbation
* ability to communicate and read Norwegian

Exclusion Criteria:

* parents of children with chronic diseases who have direct access to the acute ward, children with oxygen saturation less than 90 %, or other very sick children who need urgent treatment

Ages: 10 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
parental anxiety | at discharge from the acute ward. An average stay in the acute ward is about 5 hours.
  evaluated with the State-Trait Anxiety Inventory (STAI) (translated to Norwegian)

SECONDARY OUTCOMES:
parental satisfaction with nursing care | at discharge from the acute ward. An average stay in the acute ward is about 5 hours.
  evaluated with the Consumer Emergency Care Satisfaction Scale (CECSS)
Parental satisfaction with the health information given in the acute ward. | 1-2 weeks after discharge from the hospital. An average stay in the acute ward is about 5 hours, and an average stay in the children's department is 2 days.
  Evaluated with a structured telephone interview 1-2 weeks after hospital discharge, performed by the main researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Skranes, MD, PhD, Study Director — Norwegian University of Science and Technology; Henrik Døllner, MD, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- Department of Pediatrics, St. Olav's University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Botngard A, Skranes LP, Skranes J, Dollner H. Multimedia based health information to parents in a pediatric acute ward: a randomized controlled trial. Patient Educ Couns. 2013 Dec;93(3):389-93. doi: 10.1016/j.pec.2013.04.017. Epub 2013 May 15. PMID 23684375
- See also: an open online resource in Norwegian for parents of small children, containing videos, audio clips, animations, illustrations, pictures and text materials regarding children's illnesses and normal development — http://www.syktbarn.no
- See also: an open online resource for parents of small children, containing videos, audio clips, animations, illustrations, pictures and text materials regarding children's illnesses and normal development — http://www.childhealthguide.com